CLINICAL TRIAL: NCT04695158
Title: Determination of Hemoglobin A1c, Lipid Profiles, Homocysteine, Oxidative Stress Parameters and Physical Activity Levels in Patients With Type II Diabetes and/or COVID-19
Brief Title: Blood Sample Measurements and Physical Activity Levels in Type II Diabetes and/or COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Izmir Bakircay University (Other)
Collaborators: Cigli Regional Training Hospital (Other); Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Kadirhan Ozdemir, PT, PhD., Assist. Prof., Izmir Bakircay University
Other Study IDs: 2020-12-143
Record Dates: First submitted 2021-01-02; First posted 2021-01-05 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Diabetes Mellitus, Type 2
Keywords: Hemoglobin A1c; Lipid profiles; Homocystein; Oxidative stress parameters; Physical activity level; Covid19 (SARS-CoV-2); Type II Diabetes Mellitus
MeSH Terms: conditions — COVID-19; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 group (Group I): Patients diagnosed with COVID-19 will be in this group. No additional intervention will be applied in this group except the routine COVID-19 treatment according to the Adult Patient Treatment Guide which published by the Ministry of Health, Republic of Turkey on 9 October 2020.
  Interventions: Drug: COVID-19 group (Group I)
- Type II Diabetes Mellitus and COVID-19 group (Group II): Patients diagnosed with both Type II Diabetes Mellitus and COVID-19 will be in this group. No additional intervention will be applied in this group except the routine COVID-19 treatments according to the Adult Patient Treatment Guide which published by the Ministry of Health, Republic of Turkey on 9 October 2020 and routine treatment for Type II Diabetes Mellitus.
  Interventions: Drug: Type II Diabetes Mellitus and COVID-19 group (Group II)
- Control group (Group III): Healthy volunteers will be in this group. No intervention will be applied in this group.

INTERVENTIONS:
Drug: COVID-19 group (Group I) — Routine COVID-19 treatment
  Groups: COVID-19 group (Group I)
Drug: Type II Diabetes Mellitus and COVID-19 group (Group II) — Routine Type II Diabetes Mellitus and COVID-19 treatments
  Groups: Type II Diabetes Mellitus and COVID-19 group (Group II)

SUMMARY:
It is known that COVID-19 has a more negative clinical course and causes higher degrees of morbidity and mortality in case of COVID-19 in diabetic patients. However, the contribution of COVID-19 to hyperglycemia and its effect on glycemic parameters are uncertain. However, it is important to investigate homocysteine and lipid profile levels, respectively, and free radical levels known to be effective in the development of cardiovascular disease and diabetes due to oxidative stress, which can provide information about the identification and diagnosis of cardiovascular complications in the COVID-19 pandemic. In addition, as the decrease in physical activity levels of individuals in the COVID-19 pandemic may cause possible secondary complications such as an increase in the risk of cardiovascular disease, determining the physical activity levels of individuals and encouraging them to physical activity is another important parameter to minimize the negative effects of the process. Patients who applied to Izmir Bakircay University Cigli Training and Research Hospital (Cigli Regional Education Hospital) and hospitalized in the COVID-19 service and healthy controls are planning to include in this study. Patients diagnosed with COVID-19 will be included in Group I (n: 20), patients diagnosed with both Type II Diabetes Mellitus and COVID-19 will be included in Group II (n: 20) and healthy controls will be included in Group III (n:20). Hemoglobin A1c levels, lipid profiles, homocysteine, free radical levels and physical activity levels will be compared between groups. In addition, the change in the relevant variables before and after COVID-19 treatment will be determined by in-group comparisons in Group I and Group II. This study, which has a prospective and randomized controlled research plan, is planned to be carried out between January and February 2021. Research data will be obtained from blood samples taken from participants. In addition, data on physical activity levels will be collected through a questionnaire. After analyzing the data obtained from the research with appropriate statistical methods, the data will be evaluated.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) pandemic caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) results in significantly higher morbidity and mortality in patients with concomitant diseases such as diabetes mellitus and hypertension.

Glycemic management is of much more interest for both diabetes and COVID-19 patients, as diabetes has been reported to be associated with the poor prognosis of COVID-19. There is evidence that better glycemic control in COVID-19 patients is closely related to improved clinical outcomes. However, whether COVID-19 contributes to hyperglycemia is confusing. It remains unclear regarding the impact of COVID-19 infection on glycemic parameters, including blood glucose and hemoglobin A1c (HbA1c).

Lipid profile assessment is an important tool that helps diagnose cardiovascular diseases. Therefore, the stability of the samples is crucial for the analysis of total cholesterol (TC), low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C) and triglycerides (TG).Stability is the ability of analyte concentrations to be minimally affected within an acceptable range over a period of time.

High plasma homocysteine levels significantly increase the incidence of vascular damage in both small and large vessels. Concentrations above the 90th percentile are associated with an increased risk of degenerative and atherosclerotic processes in the coronary, cerebral and peripheral circulatory systems. Although homocysteine is an effective cardiovascular risk biomarker and is critical for cardiovascular complications in hospitalized COVID-19 patients, studies on this parameter have not focused much on laboratory markers useful for clinical evaluation of COVID-19.

Free radicals are continuously formed at the active site of enzymes as intermediates in enzymatic reactions occurring during cell metabolism. Reactive oxygen species and reactive nitrogen, known as intermediates, sometimes leach from the active site of enzymes and accidentally interact with molecular oxygen and form free oxygen radicals.Lipids, proteins, enzymes, carbohydrates, and DNA can be damaged due to oxidative stress, random breaks and bonds in DNA chains may occur as a result of damage to membranes, damage to enzymes and structural proteins may result in cell death, and these phenomena may result in cancer, neurodegenerative and cardiovascular diseases, diabetes and It constitutes the molecular basis in the development of autoimmune disorders.

The general recommendation for thinking that an adult is physically active is to achieve at least 150 minutes of moderate or 75 minutes of vigorous vigorous activity per week, or an equivalent combination of both, and involving sedentary behavior, energy expenditure ≤ 1.5 metabolic equivalent (MET), while lying down, leaning, It is defined as any waking behavior practiced while sitting or standing. As the disease spreads all over the world, healthy people are asked to stay at home for a long time. As a result, COVID-19 has radically changed the determinants of both behaviors (individual, interpersonal, environmental, regional or national policies and global). Accordingly, it can be said that regular and joint activities decrease due to isolation and limitations, especially in the first weeks when the population has limited chances to find alternatives to keep active even at home, and reducing sedentary behavior during closure poses a significant challenge. Because of this situation, physical activity in the home environment is strongly encouraged by public health advocates to prevent the potential harmful effects of protective lifestyle regulations due to COVID-19 and to prevent the restrictions from causing physical inactivity.

The main aim of this study is to compare hemoglobin A1c levels, lipid profiles, homocysteine, oxidative stress parameters and physical activity levels in patients with COVID-19 and patients with both COVID-19 and Type II diabetes via healthy adults. The second aim is to compare the initial data obtained following the hospitalization of COVID-19 patients and patients with both COVID-19 and Type II diabetes, with the latest data obtained after treatment and before discharge.

ELIGIBILITY:
Inclusion Criteria:

* To voluntarily participate in the study
* To be diagnosed with both Type II diabetes and COVID-19 for Group I
* To be diagnosed with COVID-19 for Group II
* Not having any diagnosed chronic diseases for Group III

Exclusion Criteria:

* Patients who do not need hospitalization
* Patients with a diagnosis of Type I Diabetes Mellitus
* Patients diagnosed with renal failure and/or heart failure
* Being pregnant
* Body mass index over 40kg/m2

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in Group I and Group II will be included the study from Izmir Bakircay University Cigli Training and Research Hospital (Cigli Regional Training Hospital).
  Participants in Group III will be included the study from community sample.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change of the levels of Hemoglobin A1c and Lipid Profiles at baseline and discharge for Group I and Group II | At baseline and immediately before the discharge
  Hemoglobin A1c and lipid profiles will be determined by venous blood samples taken from the participants. Blood plasma Hemoglobin A1c levels will be analyzed using immunoturbidimetric method and Lipid Profiles including Total cholesterol, high density lipoprotein (HDL) cholesterol and Triglyceride levels will be analyzed by using colorimetric methods in Medical Biochemistry Laboratory. Very low-density lipoprotein (VLDL) cholesterol and low density lipoprotein (LDL) cholesterol will be calculated by the Friedewald formula. All these parameters will be studied on the Cobas Integra 800 biochemical analyzer (Roche Diagnostics, Gesellschaft mit beschränkter Haftung (GmbH), Mannheim, Germany).
The levels of Hemoglobin A1c and Lipid Profiles for Group III | At baseline
  Hemoglobin A1c and lipid profiles will be determined by venous blood samples taken from the participants. Blood plasma Hemoglobin A1c levels will be analyzed using immunoturbidimetric method and Lipid Profiles including Total cholesterol, HDL-C and Triglyceride levels will be analyzed by using colorimetric methods in Medical Biochemistry Laboratory. VLDL-C and LDL-C will be calculated by the Friedewald formula. All these parameters will be studied on the Cobas Integra 800 biochemical analyzer (Roche Diagnostics, GmbH, Mannheim, Germany).
Change of the levels of Homocystein and Oxidative Stress Parameters at baseline and discharge for Group I and Group II | At baseline and immediately before the discharge
  Homocystein levels will be studied by using Enzyme Chemiluminescence Immunoassay (ECLIA), and Oxidative Stress Parameters including Superoxide Dismutase (SOD), Malondialdehyde (MDA), Total Antioxidant Level (TAL) / Total Oxidant Level (TOL) will be studied by photometric method in Medical Biochemistry Laboratory.
The levels of Homocystein and Oxidative Stress Parameters for Group III | At baseline
  Homocystein levels will be studied by using Enzyme Chemiluminescence Immunoassay (ECLIA), and Oxidative Stress Parameters including Superoxide Dismutase (SOD), Malondialdehyde (MDA), Total Antioxidant Level (TAL) / Total Oxidant Level (TOL) will be studied by photometric method in Medical Biochemistry Laboratory.
Change of Physical Activity Level at baseline and discharge for Group I and Group II | At baseline and immediately after the recovery
  International Physical Activity Questionnaire-Short Form (IPAQ-SF) will be used to determine the level of physical activity for last 7 days. This questionnaire consists of 7 questions and provides information about sitting, walking, moderate activities and time spent on vigorous activities. The calculation of the total score includes the total duration and frequency of walking, moderate activity, and vigorous activity. The sitting score is calculated separately. In the evaluation of all activities, the criterion is that each activity should be done at least 10 minutes. The walking time will be multiplied by 3.3 MET (The metabolic equivalent of task) in the calculation of the walking score. In the calculation, 4 METs for moderate activity and 8 METs for vigorous activity will be taken. Physical activity levels will categorize as inactivity (<600 MET-min/week), low physical activity (600-3000 MET-min/week) and adequate physical activity (>3000 MET-min/week) minutes/week).
Physical Activity Level for Group III | At baseline and immediately after the recovery
  International Physical Activity Questionnaire-Short Form (IPAQ-SF) will be used to determine the level of physical activity for last 7 days. This questionnaire consists of 7 questions and provides information about sitting, walking, moderate activities and time spent on vigorous activities. The calculation of the total score includes the total duration and frequency of walking, moderate activity, and vigorous activity. The sitting score is calculated separately. In the evaluation of all activities, the criterion is that each activity should be done at least 10 minutes. The walking time will be multiplied by 3.3 MET (The metabolic equivalent of task) in the calculation of the walking score. In the calculation, 4 METs for moderate activity and 8 METs for vigorous activity will be taken. Physical activity levels will categorize as inactivity (<600 MET-min/week), low physical activity (600-3000 MET-min/week) and adequate physical activity (>3000 MET-min/week) minutes/week).

SECONDARY OUTCOMES:
Change of the levels of Routine Blood Samples at baseline and discharge for Group I and Group II | At baseline and immediately before the discharge
  Hemogram, levels of vitamin D, Troponin T, D-Dimer, iron, ferritin, C-reactive protein (CRP), lymphocyte/CRP ratio, neutrophil/lymphocyte ratio, levels of procalcitonin, uric acid, chlorine, blood urea nitrogen (BUN) creatine, albumin and bilirubin will be taken from patient files.
The levels of Routine Blood Samples for Group III | At baseline
  Hemogram, levels of vitamin D, Troponin T, D-Dimer, iron, ferritin, C-reactive protein (CRP), lymphocyte/CRP ratio, neutrophil/lymphocyte ratio, levels of procalcitonin, uric acid, chlorine, BUN creatine, albumin and bilirubin will be requested to be studied by the attending physician.

CONTACTS AND LOCATIONS:
Locations (1):
- Kadirhan Ozdemir, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Adult Patient Treatment Guide for COVID-19 (Ministry of Health, Republic of Turkey) — https://covid19.saglik.gov.tr/TR-66926/eriskin-hasta-tedavisi.html